CLINICAL TRIAL: NCT01677832
Title: Neuronal Correlates of Executive Functions and Self-Regulation Among Children and Adolescents With and Without ADHD in Germany and Taiwan
Brief Title: Executive Functions and Self-Regulation Among Children With and Without ADHD in Germany and Taiwan
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Collaborators: National Health Research Institutes, Taiwan (Other)
Responsible Party: Principal Investigator, Statistical Center, NTUHCTC, Susan Shur-Fen Gau, National Taiwan University Hospital
Other Study IDs: 201201062RIB
Record Dates: First submitted 2012-08-30; First posted 2012-09-03 (Estimated); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Attention-Deficit/Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- ADHD/Taiwan
- Control/Taiwan
- ADHD/Germany
- Control/Germany

SUMMARY:
Children and adolescents with ADHD are impulsive and have difficulties in regulating their behaviors. It has been suggested that a core deficit in inhibitory control may account for dysfunctional behaviors associated with this disorder. Previous research has shown that medication and the self-regulation strategy of making implementation intentions (i.e., if-then plans) are effective in enhancing children's inhibitory control, which is reflected in the behavioral as well as electrophysiological (e.g., Electroencephalogram; EEG) data on a Go/NoGo task in children with ADHD. As suggested by earlier research, however, forming implementation intentions may have different effects on people who are embedded in different cultures.

The aim of the present study is to compare the effects of medication and the self-regulation of forming implementation intentions by assessing the behavioral performance and corresponding brain activity during a Go/NoGo task in children and adolescents with and without ADHD under two different cultural contexts. Further, this study also aims at investigating the potential moderating effects of culture on making if-then plans. More important, as we know, this will be the first study to compare the effectiveness of forming implementation intentions on children and adolescents with ADHD in a cross-cultural way, which is meaningful for researchers to explore the degree of its application and expected to provide clinical psychologists an alternative perspective for ADHD treatment in the near future.

DETAILED DESCRIPTION:
For a deeper understanding of the mechanism underlying the effects of MPH and implementation intentions, neurophysiological data (with a special interest on the P300 component) during a Go/NoGo task will be assessed additionally to the behavioral performance (i.e., response times and error rates). Meanwhile, the information may contribute to a better understanding of a potential influence of culture on the effect of implementation intentions. The effect may be equally effective in the cultures, but the underlying processes might still differ. On the other hand, differences between the two cultural groups might be explained by different neurophysiological activity during the tasks.

Two primary research questions arise: (1) Are MPH and implementation intentions (i.e., if-then plans) effective in enhancing the performance of executive function tasks measured by the Go/NoGo task in children and adolescents with ADHD compared with those without ADHD within each culture? (2) Does culture play a role in moderating the effect of implementation intentions on executive function tasks in children and adolescents with ADHD, respectively? Based on the research questions, two hypotheses are formulated. First, after the treatment of MPH and the self-regulation strategy of forming implementation intentions, it would result in less inhibition errors and more increased amplitudes of NoGo P300 and NoGominusGo P300 in children and adolescents with ADHD. Second, participants with ADHD in Taiwan may benefit more from the self-regulation strategy, which is reflected in more increased amplitudes of NoGo P300 and NoGominusGo P300 than found in their counterparts in Germany. However, since this is the first study to compare the effects of forming implementation intentions in a cross-cultural way, this latter analysis is more exploratory.

ELIGIBILITY:
Inclusion Criteria:

* Participants with ADHD have to meet the criteria of ICD-10 (WHO, 1991) before enrolment.
* Participants with ADHD are diagnosed with ADHD combined subtype.
* Ages range from 10 to 14 when we conduct the study.
* IQ full score ≥ 80.

Exclusion Criteria:

* The subjects will be excluded from the study if they currently meet criteria or have a history of the following condition as defined by DSM-IV: Schizophrenia, Schizoaffective Disorder, Organic Psychosis, Mental Retardation, or Pervasive Developmental Disorder. Moreover, the subjects will be excluded from the control group if have a history of the following condition as defined by DSM-IV: ADHD or ASD in addition to the above exclusion criteria.

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Participants will be recruited respectively in Germany and Taiwan using the same standardized procedures according to the protocol. Children and adolescents with and without ADHD between the ages 10 to 14, with an IQ full score ≥ 80, will participate in this study. Participants with ADHD have to meet the criteria of ICD-10 (WHO, 1991) before enrolment. They are diagnosed with ADHD combined subtype and have no comorbid disorders. None of the controls are clinically diagnosed with any disorders and take any medication. Both samples should be matched according to the variables: gender, IQ, and socio-economic status (SES).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Shur-Fen Gau, MD, PhD, Principal Investigator — National Taiwan University Hospital & College of Medicine
Locations (1):
- National Taiwan Univeristy Hospital, Taipei, Taiwan